CLINICAL TRIAL: NCT03330899
Title: A Phase I Randomized, Double-blind, Placebo-controlled, Dose Finding Clinical Trial to Evaluate the Safety and Immunogencity of H7N9 Influenza Antigen Adjuvanted With 2 Different Adjuvant Formulations in Healthy Adult Volunteers in Brazil
Brief Title: Safety and Immunogencity of H7N9 Influenza Antigen With 2 Adjuvant Formulations in Healthy Adults in Brazil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLP-01-IB
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Influenza; H7N9 Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 15 mcg H7N9 + adjuvant IB160 (Active Comparator): Participants in this arm will receive one dose of the combination (15 mcg H7N9 antigen + adjuvant IB160) at Day 0 and another dose at Day 28.
  Each dose after combination = 0,5 ml 15 mcg of the monovalent H7N9 antigen per dose
  Interventions: Biological: H7N9 antigen + adjuvant IB160
- 7.5 mcg H7N9 + adjuvant IB160 (Active Comparator): Participants in this arm will receive one dose of the combination (7.5 mcg H7N9 antigen + adjuvant IB160) at Day 0 and another dose at Day 28.
  Each dose after combination = 0,5 ml 7.5 mcg of the monovalent H7N9 antigen per dose
  Interventions: Biological: H7N9 antigen + adjuvant IB160
- 3.75 mcg H7N9 + adjuvant IB160 (Active Comparator): Participants in this arm will receive one dose of the combination (3.75 mcg H7N9 antigen + adjuvant IB160) at Day 0 and another dose at Day 28.
  Each dose after combination = 0,5 ml 3.75 mcg of the monovalent H7N9 antigen per dose
  Interventions: Biological: H7N9 antigen + adjuvant IB160
- 15 mcg H7N9 + adjuvant SE (Active Comparator): Participants in this arm will receive one dose of the combination (15 mcg H7N9 antigen + adjuvant SE) at Day 0 and another dose at Day 28.
  Each dose after combination = 0,5 ml 15 mcg of the monovalent H7N9 antigen per dose
  Interventions: Biological: H7N9 antigen + adjuvant SE
- 7.5 mcg H7N9 + adjuvant SE (Active Comparator): Participants in this arm will receive one dose of the combination (7.5 mcg H7N9 antigen + adjuvant SE) at Day 0 and another dose at Day 28.
  Each dose after combination = 0,5 ml 7.5 mcg of the monovalent H7N9 antigen per dose
  Interventions: Biological: H7N9 antigen + adjuvant SE
- 3.75 mcg H7N9 + adjuvant SE (Active Comparator): Participants in this arm will receive one dose of the combination (3.75 mcg H7N9 antigen + adjuvant SE) at Day 0 and another dose at Day 28.
  Each dose after combination = 0,5 ml 3.75 mcg of the monovalent H7N9 antigen per dose
  Interventions: Biological: H7N9 antigen + adjuvant SE
- 15 mcg H7N9 without adjuvant (Active Comparator): Participants in this arm will receive one dose of the 15 mcg H7N9 antigen without adjuvant at Day 0 and another dose at Day 28.
  Each dose = 0,5 ml
  Interventions: Biological: H7N9 antigen without adjuvant
- Placebo (PBS) (Placebo Comparator): Participants in this arm will receive one dose of Placebo (PBS) at Day 0 and another dose at Day 28.
  Each dose = 0,5 ml
  Interventions: Biological: Placebo (PBS)

INTERVENTIONS:
Biological: H7N9 antigen + adjuvant IB160 — H7N9 monovalent (fragmented and inactivated)
  Arms: 15 mcg H7N9 + adjuvant IB160; 3.75 mcg H7N9 + adjuvant IB160; 7.5 mcg H7N9 + adjuvant IB160
Biological: H7N9 antigen + adjuvant SE — H7N9 monovalent (fragmented and inactivated)
  Arms: 15 mcg H7N9 + adjuvant SE; 3.75 mcg H7N9 + adjuvant SE; 7.5 mcg H7N9 + adjuvant SE
Biological: H7N9 antigen without adjuvant — H7N9 monovalent (fragmented and inactivated)
  Arms: 15 mcg H7N9 without adjuvant
Biological: Placebo (PBS) — Placebo (Phosphate Buffered Saline -PBS)
  Arms: Placebo (PBS)

SUMMARY:
The overall aim of this study is to evaluate the safety, immunogenicity and dose sparing effects of H7N9 influenza antigen formulated with 2 different adjuvants .

DETAILED DESCRIPTION:
Following the emergence of avian influenza A/H7N9 influenza virus in humans in China in March 2013, the WHO Essential Regulatory Laboratories prepared candidate vaccine viruses and reagents for further development and several manufacturers have developed various inactivated influenza vaccines with and without adjuvant against A/H7N9 and tested these candidates in trials in healthy adults. The overall aim of this study is to evaluate the safety, immunogenicity and dose sparing effects of H7N9 influenza antigen produced by Butantan Institute in combination with 2 different adjuvants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female (non-pregnant) adults 18 through 59 years of age at the enrollment visit.
* To be available to participate in the study throughout its duration (approximately seven months).
* Healthy, as established by the medical history, physical examination, and screening laboratory evaluations.
* Capable and willing to complete Participant Diaries and willing to return for all follow-up visits.
* To demonstrate intention to participate in the study, as documented by signature in the study´s informed consent form.
* For females of child-bearing potential, willing to utilize reliable birth control measures from Day 0 through at least 60 days following the last study vaccination.

Exclusion Criteria:

* Participation in another clinical trial involving any experimental therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Evidence of active neurological, cardiac, pulmonary, hepatic or renal disease as clinical history and/or physical examination (except hypertension under control).
* Compromised immune system diseases including: HIV, Hepattis B and C, diabetes mellitus, cancer (except basal cell carcinoma) and autoimmune diseases.
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements.
* Abusive usage of alcohol or drugs in the past 12 months that has caused medical, professional or family problems, indicated by clinical history.
* Known systemic hypersensitivity to eggs or to any component of the vaccine.
* History of severe adverse reaction after previous administration of an Influenza vaccine within 6 weeks following vaccination.
* History of Guillain-Barre Syndrome or other demyelinating disease.
* Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
* Diagnosis of asthma with a history of hospitalization related to this condition in the last six months due to illness.
* Suspected or confirmed fever in the 3 days prior to vaccination or axillary temperature greater than 37.8 ° C on the day of vaccination.
* Use of corticosteroids (except topical or nasal) or other immunosuppressive drugs within 42 days before study initiation/baseline. It will be considered immunosuppressive dose of corticosteroids the equivalent to a dose ≥10 mg of prednisone per day for over 14 days.
* Impaired coagulation due to chronic disease or due to use anticoagulant medication (warfarin or heparin) in the 7 days preceding vaccination.
* Have received live virus vaccine within 28 days or killed virus vaccine in the last 14 days prior to vaccination, or have a scheduled immunization from the first study vaccination until 21 days after the second vaccination.
* Have received any influenza A/H7 vaccine.
* History of asplenia.
* Have received blood products in the past 6 months, including transfusions or immunoglobulin, or scheduled administration of blood products or immunoglobulin for the first 21 days after vaccination.
* Any other condition that might put at risk the safety/rights of a potential participant or his/her compliance with this protocol in investigator's opinion or his representative physician.
* Laboratory values at screening equal to or greater than Grade 2 will be considered to be exclusionary. Vital signs may be performed up to three times to allow for transient conditions to resolve. Screening laboratory values that are out of range, but are considered to be due to an acute illness or process may be repeated once. Grade 1 laboratory values will be reviewed by a licensed study clinician and the clinician will determine whether the laboratory abnormality is clinically significant and should be considered exclusionary. If determined to be clinically insignificant, the study team is not required to follow the laboratory until resolution or the value is determined to be clinically stable.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 432 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with solicited local Adverse Events over the 7-day period post each study injection. | 7-day period post each study injection (Days 0-6)
  Solicited local Adverse Events (AE) include erythema, swelling/induration, pain/tenderness, ecchymosis, pruritis.
  The participant will be given a Participant Diary, a digital thermometer and ruler in which the participant will be asked to record any local and/or systemic reactions.
  The participant will have been instructed that if he/she experiences an AE requiring medical care, the participant should inform the study staff as soon as possible and seek medical care as appropriate.
  A visit will be schedule to occur 7 days after each study injection. Study staff will review the Participant Diary and interim history with the participant and inquire about new medical events, which will be recorded in the appropriate Clinical Research Forms.
Number of participants with solicited systemic Adverse Effects over the 7-day period post each study injection. | 7-day period post each study injection (Days 0-6)
  Solicited systemic Adverse Events (AE) include fever, fatigue/malaise, myalgia, arthralgia, chills, nausea/vomiting, and headache.
  The participant will be given a Participant Diary, a digital thermometer and ruler in which the participant will be asked to record any local and/or systemic reactions.
  The participant will have been instructed that if he/she experiences an AE requiring medical care, the participant should inform the study staff as soon as possible and seek medical care as appropriate.
  A visit will be schedule to occur 7 days after each study injection. Study staff will review the Participant Diary and interim history with the participant and inquire about new medical events, which will be recorded in the appropriate Clinical Research Forms.
Number of participants with unsolicited local and/or systemic Adverse Events over the 7-day period post each study injection. | 7-day period post each study injection (Days 0-6)
  Unsolicited local and/or systemic Adverse Events include any AE not include in the description of solicited AE, as described in Outcome 1 and 2.
  The participant will be given a Participant Diary, a digital thermometer and ruler in which the participant will be asked to record any local and/or systemic reactions.
  The participant will have been instructed that if he/she experiences an AE requiring medical care, the participant should inform the study staff as soon as possible and seek medical care as appropriate.
  A visit will be schedule to occur 7 days after each study injection. Study staff will review the Participant Diary and interim history with the participant and inquire about new medical events, which will be recorded in the appropriate Clinical Research Forms.

SECONDARY OUTCOMES:
Number of participants with unsolicited local and/or systemic Adverse Events over the 28-day period post each study injection. | 28-day period post each study injection (Days 0-27)
  Unsolicited local and/or systemic Adverse Events include any AE not include in the description of solicited AE, as described in Outcome 1 and 2.
  A visit will be schedule to occur 28 days after each study injection. Study staff will review the Participant Diary and interim history with the participant and inquire about new medical events, which will be recorded in the appropriate Clinical Research Forms.
Number of participants with Serious Adverse Events over the 222-day period post second study injection. | 222-day period post the second study injection (Days 0-221)
  Serious Adverse Event (SAE) is defined as an adverse event that meets one of the following conditions:
  * Death.
  * Life-threatening.
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
  * Results in congenital anomaly/birth defect.
  * Results in a persistent or significant disability or incapacity.
  * Important medical events that might not result in death, be life-threatening, or require hospitalization might be considered SAEs when, based upon appropriate medical judgment, the event might jeopardize the well-being of the participant and require medical or surgical intervention to prevent one of the outcomes listed above.
  Participants will be contacted by phone on Day 222 after administration of second dose of study product for (a) closure of any ongoing AEs and concomitant medications; and (b) collection of any SAEs and new concomitant medications, if associated with the SAE reported.
Number of participants that presented seroconversion at day 28, 45 and 56 post first study injection | 56-day period post the first study injection
  Seroconvertion is defined as: prevaccination Hemagglutination-inhibition test (HI) antibody titer ≤1:10 and postvaccination HI antibody titer ≥1:40, or prevaccination HI antibody titer ≥1:10 and a postvaccination increase by a factor of four or more).
  Participants will be invited to return on days 28, 45 and 56 post first study injection, when blood samples will be taken for HI testing.
Number of participants that presented seroprotection at day 28, 45 and 56 post first study injection | 56-day period post the first study injection
  Seroprotection is defined as postvaccination Hemagglutination-inhibition test (HI) antibody titer ≥ 1:40.
  Participants will be invited to return on days 28, 45 and 56 post first study injection, when blood samples will be taken for HI testing.
Geometric mean of Hemagglutination-inhibition titre at day 28, 45 and 56 post first study injection | 56-day period post the first study injection
  Geometric mean of Hemagglutination-inhibition test titre will be calculated for the different groups of participants at day 28, 45 and 56 post first study injection.
  Participants will be invited to return on days 28, 45 and 56 post first study injection, when blood samples will be taken for HI testing.

CONTACTS AND LOCATIONS:
Overall Officials: Esper Kallas, PhD, Principal Investigator — University of Sao Paulo
Locations (3):
- Brazil (3):
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Centro de Pesquisas Clínicas do Instituto Central do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Centro de Pesquisa Clínica do Instituto da Criança do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - ICr/HCFMUSP, São Paulo, São Paulo

REFERENCES:
- [Derived] Vanni T, Thome BC, Sparrow E, Friede M, Fox CB, Beckmann AM, Huynh C, Mondini G, Silveira DH, Viscondi JYK, Braga PE, Silva AD, Salomao MDG, Piorelli RO, Santos JP, Gattas VL, Lucchesi MBB, Oliveira MMM, Koike ME, Kallas EG, Campos LMA, Coelho EB, Siqueira MAM, Garcia CC, Miranda MD, Paiva TM, Timenetsky MDCST, Adami EA, Akamatsu MA, Ho PL, Precioso AR. Dose-sparing effect of two adjuvant formulations with a pandemic influenza A/H7N9 vaccine: A randomized, double-blind, placebo-controlled, phase 1 clinical trial. PLoS One. 2022 Oct 18;17(10):e0274943. doi: 10.1371/journal.pone.0274943. eCollection 2022. PMID 36256646